CLINICAL TRIAL: NCT04511234
Title: Randomized Controlled Trial of First Sirolimus Coated Balloon Versus Standard Balloon Angioplasty in The Treatment of Superficial Femoral Artery and Popliteal Artery Disease
Brief Title: Sirolimus Coated Balloon Versus Standard Balloon for SFA and Popliteal Artery Disease
Acronym: FUTURE-SFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concept Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FUTURE SFA
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Artery Disease; Atherosclerosis; Arterial Disease
Keywords: PAD; DCB; PTA; Sirolimus
MeSH Terms: conditions — Peripheral Arterial Disease; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomised via a secure online system to a labelled device and to receive either Magic Touch sirolimus drug coated balloon in addition to standard balloon angioplasty or standard balloon angioplasty and placebo balloon.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MagicTouch PTA sirolimus drug coated balloon (DCB) (Experimental): MagicTouch PTA sirolimus drug coated balloon (DCB) in addition to standard balloon angioplasty
  Interventions: Device: MagicTouch PTA sirolimus drug coated balloon (DCB)
- Placebo balloon angioplasty (Active Comparator): Placebo balloon angioplasty in addition to standard balloon angioplasty (PTA)
  Interventions: Device: POBA standard balloon

INTERVENTIONS:
Device: MagicTouch PTA sirolimus drug coated balloon (DCB) — For participants randomised to MagicTouch PTA sirolimus DCB, following successful plain balloon angioplasty of the arterial lesion, (defined as <30% residual stenosis after treatment at rated burst pressure of the angioplasty balloon), MagicTouch PTA sirolimus coated balloon will be applied at the lesion after appropriate sizing using the diameter of the plain balloon angioplasty.
  Arms: MagicTouch PTA sirolimus drug coated balloon (DCB)
Device: POBA standard balloon — For participants randomised to the standard balloon angioplasty group, a placebo standard balloon which is identical to the SCB will also be applied at the lesion after appropriate sizing using the diameter of the plain balloon angioplasty.
  Arms: Placebo balloon angioplasty

SUMMARY:
This study aims to conduct a randomized, double blind, randomised controlled multicentre trial of sirolimus drug coated balloon versus standard percutaneous transluminal angioplasty for the treatment of superficial and popliteal arterial disease.

DETAILED DESCRIPTION:
The burden of limb loss as a result of peripheral arterial disease (PAD) is high and this problem is set to worsen globally. Treatment of PAD primarily involves revascularisation of the limb. Angioplasty as a first line strategy of revascularization over surgical procedures has been adopted by most vascular centers. Local drug delivery using drug coated balloons (DCB) during angioplasty for PAD can successfully deliver effective local tissue concentrations of anti-proliferative drugs to the lesions in the artery involved in the PAD. This offers the potential for sustained anti-restenotic efficacy.

Randomized trials have shown superiority of Paclitaxel DCBs over just plain-balloon angioplasty for treatment of PAD, and DCB is now considered the standard of care. However a recent meta-analyses which showed increased mortality at two years in patients treated with paclitaxel DCBs have called into question the safety of paclitaxel based DCBs.

Alternative drugs for DCBs are therefore urgently needed and sirolimus offers an attractive alternative. Compared to Paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety. It has a high transfer rate to the vessel wall and has been shown to effectively inhibit neointimal hyperplasia in the porcine coronary model. In the coronary artery interventions, preliminary clinical studies using Sirolimus DCBs have also shown excellent procedural and 6 month patency.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years or minimum age
2. Rutherford class 3 to 6 in the target limb

   Intraoperative Inclusion Criteria
3. Single or sequential de novo or re-stenotic lesions (stenosis of > 50% or occlusions) from 2 to 20cm in the femoropopliteal arteries. Lesion is considered as one lesion if there is maximum of 30mm gap between lesions at discretion of investigator. Femoropopliteal arteries are superficial femoral artery, popliteal artery P1 and P2
4. Inflow free from flow limiting lesions (<50% stenosis) confirmed by duplex or angiography. Subjects with flow limiting inflow lesions (>50% stenosis) can be included if lesion had been treated successfully (<30% residual stenosis) before or during the index procedure.
5. At least one non-occluded crural vessel (ie. without significant stenosis) with angiographically documented run off to the foot.

Exclusion Criteria:

1. Comorbid conditions limiting life expectancy ≤ 1 year
2. Subject is currently participating in another investigational drug or device study that has not reached first primary endpoint yet
3. Subject is pregnant or planning to become pregnant during the course of the study
4. Heel gangrene
5. Prior bypass surgery of target vessel
6. Planned amputation of the target limb
7. Previously implanted stent in the target lesion
8. Vulnerable or protected adults
9. Bleeding diathesis or another disorder such as gastrointestinal ulceration which restrict the use of clopidogrel or aspirin
10. Known allergy to sirolimus

    Intraoperative Exclusion Criteria
11. Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations)
12. Failure to obtain <30% residual stenosis in a pre-existing lesion
13. Highly calcific lesions
14. Use of DCBs, drug eluting stent, specialty balloons or artherectomy devices during the index procedure. (Non-compliant balloons are not considered specialty balloons)
15. Lesions requiring retrograde access (SAFARI)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency at 6 months | 6 Months
  Primary patency rate at 6 months defined as proportion of subjects with duplex ultrasonography-derived peak systolic velocity ratio of < 2.4 (in absence of target lesion revascularisation)

SECONDARY OUTCOMES:
Device and procedure related death | 1, 6, 12 and 24 Months
  Proportion of device and procedure related death
All-cause death | 1, 6, 12 and 24 Months
  Proportion of subjects died by any cause
Major target limb amputation | 1, 6, 12 and 24 Months
  Proportion of major target limb amputation
Target vessel thrombosis | From day 0 to day 14
  Proportion of subjects with target vessel thrombosis
Proportion of subjects who experienced either death at 6 month or major target limb amputation at 6 month or target vessel thrombosis within 14 days | Day 0 to day 14, 6 Months
  Proportion of subjects who experienced either death at 6 month or major target limb amputation at 6 month or target vessel thrombosis within 14 days
Occurrence of adverse events (AEs), serious AEs and AEs related to device and Occurrence of adverse events (AEs), serious AEs and AEs related to device and procedure | From Day 0 to 24 Months Follow-up
  Occurrence of adverse events (AEs), serious AEs and AEs related to device and Occurrence of adverse events (AEs), serious AEs and AEs related to device and procedure
Procedural Success | From Day 1 to discharge up to maximum of 30 days
  Proportion of subjects with procedural success during hospital stay
Proportion of subjects who are free from clinically-driven Target Lesion Revascularization (TLR) | 6,12 and 24 Months
  Proportion of subjects who are free from clinically-driven TLR
Proportion of subjects who are free from clinically-driven Target Vessel Revascularization (TVR) | 6,12 and 24 Months
  Proportion of subjects who are free from clinically-driven Target Vessel Revascularization (TVR)
Primary patency | 12 and 24 Months
  Primary patency rate at 12 and 24 months
Restenosis | 6, 12 and 24 Months
  Proportion of subjects with restenosis
Subjects who are free from MAE | 6 Months
  Proportion of subjects who are free from MAE
Amputation-free survival | 6, 12 and 24 Months
  Amputation-free survival
Clinical Success | 6, 12 and 24 Months
  Proportion of subjects with clinical Success at 6, 12 and 24 months, Clinical success is defined as Improvement in Rutherford classification compared to the pre-procedure Rutherford classification
Device success | Day 1
  Proportion of subjects with device success at day 1
Technical success | Day 1
  Proportion of subjects with technical success at day 1
Wound assessment (if any) | 1, 6, 12, 24 Months
  Wound assessment (if any)
Toe Pressure or ABPI assessment | 6, 12, 24 Months
  Toe Pressure or ABPI assessment

OTHER OUTCOMES:
Improvement of quality of life | 12 and 24 months
  Mean change from baseline in EuroQol-5Dimensions (EQ-5D) health-related quality of life questionnaire score at 12 and 24 months. The score ranges from 0 to 1, and a higher score means a better outcome
Walking impairment | 12 and 24 months
  Mean change from baseline in walking impairment questionnaire score at 12 and 24 months. The score ranges form 0% t 100%, and a higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Edward Choke, Principal Investigator — Sengkang General Hospital
Locations (20):
- Singapore (6):
  - Khoo Teck Puat Hospital, Singapore
  - National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaoshiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Tzuchi Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (6):
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Vajira Hospital, Bangkok
  - Thammasat University Hospital, Pathum Thani

REFERENCES:
- [Background] Giacoppo D, Cassese S, Harada Y, Colleran R, Michel J, Fusaro M, Kastrati A, Byrne RA. Drug-Coated Balloon Versus Plain Balloon Angioplasty for the Treatment of Femoropopliteal Artery Disease: An Updated Systematic Review and Meta-Analysis of Randomized Clinical Trials. JACC Cardiovasc Interv. 2016 Aug 22;9(16):1731-42. doi: 10.1016/j.jcin.2016.06.008. PMID 27539695
- [Background] Clever YP, Peters D, Calisse J, Bettink S, Berg MC, Sperling C, Stoever M, Cremers B, Kelsch B, Bohm M, Speck U, Scheller B. Novel Sirolimus-Coated Balloon Catheter: In Vivo Evaluation in a Porcine Coronary Model. Circ Cardiovasc Interv. 2016 Apr;9(4):e003543. doi: 10.1161/CIRCINTERVENTIONS.115.003543. PMID 27069105
- [Background] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764